CLINICAL TRIAL: NCT06412588
Title: Dual Therapy With Vonoprazan Plus Amoxicillin or Doxycycline Versus Bismuth Quadruple Therapy for Helicobacter Pylori Eradication:A Prospective, Multicenter, Open-label Randomized Controlled Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Zhang, Director of Gastroenterology, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20240123-18
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori Infection; Dual therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A Bismuth quadruple (Active Comparator): Vonoprazan 20 mg, bid + amoxicillin 1.0 g, bid + doxycycline 0.1 g, bid + bismuth, treatment course 14 days
  Interventions: Drug: Vonoprazan+amoxicillin+doxycycline+bismuth for 14 days
- Group B Amoxicillin Dual therapy (Experimental): Vonoprazan 20 mg, bid + amoxicillin 1.0 g, bid , treatment course 14 days
  Interventions: Drug: Vonoprazan+Amoxicillin
- Group C doxycycline Dual therapy (Experimental): Vonoprazan 20 mg, bid +doxycycline 0.1 g, bid，treatment course 14 days
  Interventions: Drug: Vonoprazan+doxycycline

INTERVENTIONS:
Drug: Vonoprazan+amoxicillin+doxycycline+bismuth for 14 days — Group A:The patient was treated with oral Vonoprazan 20 mg, bid + amoxicillin 1.0 g, bid + doxycycline 0.1 g, bid + bismuth for 14 days.
  Other Names: Doxycycline-based Bismuth Quadruple Therapy
  Arms: Group A Bismuth quadruple
Drug: Vonoprazan+Amoxicillin — Group B: Patients were treated with oral Vonoprazan 20mg, bid + amoxicillin 1.0g, bid for 14 days.
  Other Names: Vonoprazan+Amoxicillin Dual therapy
  Arms: Group B Amoxicillin Dual therapy
Drug: Vonoprazan+doxycycline — Group C: Patients were treated with oral Vonoprazan 20 mg, bid + doxycycline 0.1 g, bid for 14 days.
  Other Names: Vonoprazan+doxycycline Dual therapy
  Arms: Group C doxycycline Dual therapy

SUMMARY:
It is planned to select Hp infection patients in a number of tertiary hospitals in Jiangsu and randomly divide them into three groups: group A is the classic group, receiving Vonoprazan 20mg, bid + amoxicillin 1.0g, bid + doxycycline 0.1g, bid + colloidal pectin bismuth 0.3g, bid and group C are double groups, respectively, receiving standard dose amoxicillin (1.0 g, bid) combined with vonorrasan dual regimen and doxycycline (0.1g, bid) combined with Vonoprazan dual regimen, the treatment course of the three groups was 14 days, and the oral dose of Vonoprazan was 20mg, bid, the eradication rate, adverse reactions, compliance and other aspects of the three groups were compared, In order to obtain a safe, efficient, economical and convenient Hp eradication program with a wider range of applications.

DETAILED DESCRIPTION:
It is planned to select Hp infection patients in a number of tertiary hospitals in Jiangsu and randomly divide them into three groups: group A is the classic group, receiving Vonoprazan 20mg, bid + amoxicillin 1.0g, bid + doxycycline 0.1g, bid + colloidal pectin bismuth 0.3g, bid and group C are double groups, respectively, receiving standard dose amoxicillin (1.0 g, bid) combined with vonorrasan dual regimen and doxycycline (0.1g, bid) combined with vonorrasan dual regimen, the treatment course of the three groups was 14 days, and the oral dose of Vonoprazan was 20mg, bid, the eradication rate, adverse reactions, compliance and other aspects of the three groups were compared, In order to obtain a safe, efficient, economical and convenient Hp eradication program with a wider range of applications.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old;
2. Patients confirmed to be positive for H. pylori by 13C-UBT or 14C-UBT;
3. Patients who have not received Helicobacter pylori eradication therapy before, or patients who have failed to eradicate in the early stage but have not received eradication therapy within half a year;
4. Voluntarily join this trial and sign the informed consent form.

Exclusion Criteria:

1. Allergy to the study drug (penicillin, amoxicillin, Vonoprazan, doxycycline, etc.);
2. Patients with confirmed active peptic ulcer;
3. Patients who have received Helicobacter pylori eradication therapy within half a year;
4. Use of antibiotics, bismuth, and histamine H2 receptor antagonists or PPIs for the first 2 weeks before starting study treatment;
5. Use of adrenocorticosteroids, non-steroidal anti-inflammatory drugs, anticoagulants, barbiturates, phenytoin, or carbamazepine drugs;
6. History of esophageal or gastric surgery;
7. Pregnant or lactating women;
8. Alcoholism
9. Suffering from serious concomitant diseases, such as liver disease, cardiovascular disease, lung disease, kidney disease;
10. Hepatic insufficiency caused by hepatitis, fatty liver and other reasons;
11. Gastric mucosa-associated lymphoid tissue lymphoma (MALT), malignant tumor diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 810 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
HP eradication rate | 4-6 weeks after the end of the last dose
  The eradication effect of Helicobacter pylori was tested by 13C-UBT or 14C-UBT

SECONDARY OUTCOMES:
Patient compliance | Within 3 days after the end of treatment
  Rate of drug consumption during the treatment period of the subjects

OTHER OUTCOMES:
Security observations | Within 3 days after the end of treatment
  Adverse drug reactions

IPD SHARING:
Plan to Share IPD: No